CLINICAL TRIAL: NCT04696081
Title: Multicenter International Prospective Registry to Identify Major Cardiovascular Events Associated With the Occurrence of Atrial Fibrillation in Active Cancer Patients
Brief Title: Atrial Fibrillation in Active Cancer Patients
Acronym: AFIB-CANCER
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Marseille, France (Unknown); Hospices Civils de Lyon, France (Unknown); Centre Francois Baclesse, Caen, France (Unknown); University Hospital of Saint-Etienne, France (Unknown); Hôpital Lariboisière Fernand Widal, Paris, France (Unknown); Institut de Cancérologie de l'Ouest Nantes, France (Unknown); Fundacion Cardio Onco, Santiago, Chile (Unknown); Hunter New England Area Health Service, University of Newcastle, Australia (Unknown); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco122020
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Drug Toxicity; Atrial Fibrillation; Cardiovascular Complication
MeSH Terms: conditions — Neoplasms; Drug-Related Side Effects and Adverse Reactions; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: occurence of atrial fibrillation — all adult patients with an active cancer and experiencing atrial fibrillation will be consecutively include. Active cancers will be defined according Agnelli et al. (NEJM 2020; 382:1599-1607).

SUMMARY:
Atrial fibrillation is a common complication of both cancer and anticancer drugs but the consequences of such events remain poorly known and are not adressed in both phase III oncological trials and cardiological guidelines. The objective of this study is to create a prospective multicenter international registry of adult patients with an active cancer and experiencing atrial fibrillation to study major cardiovascular events occurrence during a 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* outpatients or hospitalized patients
* with a confirmed cancer (other than basal-cell or squamous-cell carcinoma of the skin, primary brain tumor, known intracerebral metastases, or acute leukemia) and an active cancer (defined as cancer that had been diagnosed within the past 6 months or recurrent locally advanced or metastatic cancer, for which anticancer treatment was being given at the time of enrollment or during 6 months before enrollment)
* at least 1 episode of atrial fibrillation (new onset AF occuring after cancer diagnosis or history of paroxysmal of persistant AF prior to cancer diagnosis and an AF recurrence after cancer diagnosis)
* in sinus rhythm at the time of cancer diagnosis

Exclusion Criteria:

* patient with palliative cares or other conditions resulting in short term death (death expected in the month following atrial fibrillation occurrence)
* history of long-standing persistant or permanent AF prior to cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a cancer will defined as patients with confirmed cancer other than basal-cell or squamous-cell carcinoma of the skin, primary brain tumor, known intracerebral metastases, or acute leukemia.
  Active cancer will be defined as cancer that had been diagnosed within the past 6 months or recurrent locally advanced or metastatic cancer, and an anticancer treatment given at the time of enrollment or during 6 months before enrollment (according to Agnelli et al. NEJM 2020).
  AF patients will be both patients with incident AF (first AF episode diagnosed after cancer diagnosis) and those with prevalent AF (AF recurrence occurring after cancer diagnosis and a first AF episode prior to cancer diagnosis)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of major cardiovascular events and death of any cause at 1 year | from inclusion in the registry to 1 year of follow-up
  Occurrence of death of any cause, cardiovascular death, heart failure, stroke, myocardial infarction in active cancer patients with atrial fibrillation.

SECONDARY OUTCOMES:
Occurrence of major cardiovascular events and death of any cause at 1 year in prevalent and incident AF patients | from inclusion in the registry to 1 year of follow-up
  Occurrence of death of any cause, cardiovascular death, heart failure, stroke, myocardial infarction in active cancer patients according to the AF type (prevalent or incident).
Description of the population of active cancer patients experiencing atrial fibrillation (in both prevalent and incidence AF patients). | at the inclusion in the registry
  Description of the population of active cancer patients experiencing atrial fibrillation. Active cancers will be defined according Agnelli et al. (NEJM 2020; 382:1599-1607).
Description of the management of atrial fibrillation in cancer patients (in both prevalent and incidence AF patients). | from inclusion in the registry to 1 year of follow-up
  Description of the management (anticoagulants, rhythm or rate control) of atrial fibrillation in cancer patients
Description of the population of active cancer patients having a major cardiovascular event | from inclusion in the registry to 1 year of follow-up
  Description of the population of patients having a major cardiovascular event among cancer patients experiencing atrial fibrillation
Identifying risk factors associated with major cardiovascular events and all cause mortality occurrence | from inclusion in the registry to 1 year of follow-up
  Identifying risk factors (clinical, EKG, biological, echocardiography) of major cardiovascular events and all cause mortality in cancer patients experiencing atrial fibrillation
Identifying factors associated with atrial fibrillation recurrence | from inclusion in the registry to 1 year of follow-up
  Identifying factors (clinical, EKG, biological, echocardiography) of atrial fibrillation recurrence in cancer patients
Occurrence of major and clinically relevant non-major bleedings (2005 ISTH definition) | from inclusion in the registry to 1 year of follow-up
  Occurrence of major and clinically relevant non-major bleedings in active cancer patients experiencing atrial fibrillation.
Identifying risk factors associated with major and clinically relevant non-major bleedings (2005 ISTH definition) | from inclusion in the registry to 1 year of follow-up
  Identifying risk factors (clinical, EKG, biological, echocardiography) of major and clinically relevant non-major bleedings in active cancer patients experiencing atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Alexandre, MD, PhD, Principal Investigator — Caen Normandy University Hospital, France
Locations (1):
- Alexandre, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alexandre J, Moslehi JJ, Bersell KR, Funck-Brentano C, Roden DM, Salem JE. Anticancer drug-induced cardiac rhythm disorders: Current knowledge and basic underlying mechanisms. Pharmacol Ther. 2018 Sep;189:89-103. doi: 10.1016/j.pharmthera.2018.04.009. Epub 2018 Apr 24. PMID 29698683
- [Background] Alexandre J, Salem JE, Moslehi J, Sassier M, Ropert C, Cautela J, Thuny F, Ederhy S, Cohen A, Damaj G, Vilque JP, Plane AF, Legallois D, Champ-Rigot L, Milliez P, Funck-Brentano C, Dolladille C. Identification of anticancer drugs associated with atrial fibrillation: analysis of the WHO pharmacovigilance database. Eur Heart J Cardiovasc Pharmacother. 2021 Jul 23;7(4):312-320. doi: 10.1093/ehjcvp/pvaa037. PMID 32353110